CLINICAL TRIAL: NCT00663663
Title: Efficacy of Telephone-Delivered Cognitive Behavioral Therapy for Chronic Pain
Brief Title: Telephone Intervention for Pain Study (TIPS)
Acronym: TIPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Dawn Ehde, Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 33597-G; R01HD057916-04 (NIH)
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Pain; Multiple Sclerosis; Amputation; Spinal Cord Injury
MeSH Terms: conditions — Chronic Pain; Multiple Sclerosis; Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Intervention 1 will consist of eight 60-minute sessions conducted by phone over eight weeks (1 session/week on average). Intervention 1 will include: (1) education about the role of cognitions (particularly catastrophizing) and pain beliefs (including control) in chronic pain and adjustment; (2) instruction in how to identify negative thinking and cognitive distortions about pain; (3) instruction in thought-stopping and cognitive-restructuring techniques, including challenging negative thoughts and core beliefs about pain; (4) instruction in utilization of positive coping self-statements; (5) relaxation techniques; (6) activity pacing and scheduling; (7) coping with pain flare-ups; and (8) relapse prevention/maintenance of gains. Each intervention 1 session will include a brief relaxation exercise practiced over the phone.
  Interventions: Behavioral: Telephone-Delivered Intervention 1
- 2 (Experimental): Intervention 2 will consist of eight 60-minute sessions conducted by phone over eight weeks (1 session/week on average), scheduled at times convenient for participants (including evenings and weekends if necessary). The sessions will cover a variety of topics, including the definition of chronic pain, the physiological processes underlying chronic pain, common pain-related conditions such as sleep disturbance, and the effects of chronic pain.
  Interventions: Behavioral: Telephone-Delivered Intervention 2

INTERVENTIONS:
Behavioral: Telephone-Delivered Intervention 1 — Intervention 1 will consist of eight 60-minute sessions conducted by phone over eight weeks. Intervention 1 will include: (1) education about the role of cognitions (particularly catastrophizing) and pain beliefs (including control) in chronic pain and adjustment; (2) instruction in how to identify negative thinking and cognitive distortions about pain; (3) instruction in thought-stopping and cognitive-restructuring techniques, including challenging negative thoughts and core beliefs about pain; (4) instruction in utilization of positive coping self-statements; (5) relaxation techniques; (6) activity pacing and scheduling; (7) coping with pain flare-ups; and (8) relapse prevention/maintenance of gains. Each intervention 1 session will include a brief relaxation exercise practiced over the phone.
  Arms: 1
Behavioral: Telephone-Delivered Intervention 2 — Intervention 2 will consist of eight 60-minute sessions conducted by phone over eight weeks (1 session/week on average), scheduled at times convenient for participants (including evenings and weekends if necessary). The sessions will cover a variety of topics, including the definition of chronic pain, the physiological processes underlying chronic pain, common pain-related conditions such as sleep disturbance, and the effects of chronic pain.
  Arms: 2

SUMMARY:
Treatments teaching people how to manage pain have been used to treat chronic pain in the general population. The purpose of this study is to see if these treatments delivered over the telephone can benefit persons with multiple sclerosis, spinal cord injury or an acquired amputation. Specifically, we want to determine if these treatments can help reduce the negative consequences that pain often causes in terms of a person's mood, daily activities, and enjoyment of life. We are also interested in finding out if these treatments decrease a person's pain.

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnosis of acquired amputation (AMP), multiple sclerosis (MS), or spinal cord injury (SCI) confirmed by participants' primary care physicians
* Average pain intensity in the past month of greater than 3 on 0-10 numeric rating scale;
* Pain is either worse or started since the onset of the disability;
* Pain of at least six months duration, with pain reportedly present greater than or equal to half of the days in the past six months;
* Read, write and understand English;
* Must be able to communicate over the phone (i.e., must be verbal);
* Age 18 years or older.

Exclusion Criteria:

* Cognitive impairment defined as one or more errors on the Six-Item screener (Callahan et al., 2002).
* Current or previous participation in a psychological treatment for pain (obtained via self-report).
* Current participation in a psychological treatment for any reason on a regular basis(obtained via self-report).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2009-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Average pain intensity | Four times in a 7-day period Pre-Treatment, Mid-Treatment, Post-Treatment, and Follow-up (6 and 12 months post-randomization).

SECONDARY OUTCOMES:
Physical Functioning-Brief Pain Inventory (Cleeland & Ryan, 1994) | pre-treatment, mid-treatment, post-treatment, and follow-up (6 and 12 months post-randomization).
Patient Health Questionnaire-8 (PHQ-8) (Kroenke & Spitzer, 2002) | pre-treatment, mid-treatment, post-treatment, and follow-up (6 and 12 months post-randomization).
Pain Catastrophizing Scale (Sullivan et al., 1995) | pre-treatment, mid-treatment, post-treatment, and followup (6 and 12 months post-randomization)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn M. Ehde, Ph.D, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States